CLINICAL TRIAL: NCT02680847
Title: An Open-label Study To Evaluate The Pharmacokinetics And Safety Of Alo-02 (Oxycodone Hydrochloride And Naltrexone Hydrochloride) Extended-release Capsules In Children And Adolescents 7-17 Years Of Age Who Require Opioid Analgesia
Brief Title: Safety and Pharmacokinetic Study of ALO-02 in Children Ages 7-17 With Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated on 08FEB2018. Pfizer has decided to withdraw the New Drug Application and has notified FDA. There are no efficacy or safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B4531015; ALO-02 PHASE 4 PEDIATRIC STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-01-20; First posted 2016-02-12 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Moderate-severe Pain
Keywords: Pediatric; pain indication; controlled release oxycodone
MeSH Terms: interventions — oxycodone naltrexone combination; Oxycodone; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALO-02 (Experimental): One arm, open label, active
  Interventions: Drug: ALO-02

INTERVENTIONS:
Drug: ALO-02 — Oral/Capsule, twice per day dosing; Treatment duration consists of a 1 to 4 week Conversion/Titration Phase leading to a 2 to 4 week Maintenance Treatment duration.
  Other Names: oxycodone hydrochloride/naltrexone hydrochloride

SUMMARY:
Safety and pharmacokinetics of an abuse-deterrent, extended-release formulation of oxycodone hydrochloride with a sequestered naltrexone core in children 7-17 with moderate-severe pain.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm study designed to characterize the PK and to evaluate the safety of ALO-02 in children and adolescents 7 to 17 years of age who require opioid analgesia for moderate-to-severe pain. The study consists of 4 study periods (screening, titration, maintenance, follow-up) occurring over a period of up to 9 weeks. The study will enroll approximately 140 children and adolescents with at least 100 subjects once stabilized during the titration period to complete a minimum of 2 of the 4 weeks study duration in the maintenance period to satisfy the PK endpoint. A safety follow-up visit is required at 1 week post-last dose.

ELIGIBILITY:
Inclusion Criteria:

* Children 7-17 with moderate to severe pain requiring around the clock treatment with an opioid analgesic.
* Be an experienced opioid user, defined as any subject treated with opioid therapy, equivalent or equal to > 6 mg per day of oxycodone, for a period of 3 consecutive days immediately prior to first day of dosing.

Exclusion Criteria:

* Columbia-Suicide Severity Rating Scale (C-SSRS) for suicidal ideation and behavior in past year.
* Hypersensitivity to morphine, naltrexone.
* A life expectancy (assessed by investigator) of less than 6 months or is no longer capable of taking medication orally.
* Undergone surgery within 3 days prior to the first day of dosing.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Research Center For Clinical Studies-West, Inc., Lancaster, California
  - Children's Hopsital Los Angeles, Los Angeles, California
  - Children's Hospital Of Los Angeles - University Of Southern California School Of Medicine, Los Angeles, California
  - Shriners Hospitals For Children Northern California, Sacramento, California
  - UC Davis Health Attn: Peter Trovitch, PharmD, Sacramento, California
  - University of California Davis, Sacramento, California
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences Systems, Chicago, Illinois
  - University of Illinois Hospital at the Medical Center, Chicago, Illinois
  - East Carolina University Brody School of Medicine(ECU), Greenville, North Carolina
  - Leo Jenkins Cancer Center Pharmacy, Greenville, North Carolina
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Investigational Drugs Services, Charleston, South Carolina
  - Medical University of South Carolina, Rutledge Tower, Pediatric Clinic, Charleston, South Carolina
  - Medical University of South Carolina, SCTR Research Nexus, Charleston, South Carolina
  - Road Runner Research, Ltd, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531015&StudyName=An%20Open-label%20Study%20To%20Evaluate%20The%20Pharmacokinetics%20And%20Safety%20Of%20Alo-02%20%28oxycodone%20Hydrochloride%20And%20Naltrexone%20Hydrochloride%29%20Extended-release%20Capsules%20In%20Children%20And%20Adolescents%207-17%20Years%20Of%20Age%20Who%20Require%20Opioid%20Analgesia
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531015&StudyName=An+Open-label+Study+To+Evaluate+The+Pharmacokinetics+And+Safety+Of+Alo-02+%28oxycodone++Hydrochloride+And+Naltrexone+Hydrochloride%29+Extended-release+Capsules+In+Children+And+Adolescents+7-17+Years+Of+Age+Who+Require+Opioid+Analgesia

RESULTS

PARTICIPANT FLOW:
Groups:
- ALO-02 <=20 mg: Oral ALO-02 capsules average daily dose ≤ 20 mg BID (the average daily dose is the total dose amount divided by the total treatment days)
- ALO-02 >20-40 mg: Oral ALO-02 capsules average daily dose >20-40 mg BID (the average daily dose is the total dose amount divided by the total treatment days)
- ALO-02 >40-80 mg: Oral ALO-02 capsules average daily dose > 40-80 mg BID (the average daily dose is the total dose amount divided by the total treatment days)
Period: Overall Study
Arm/Group | ALO-02 <=20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Started | 16 | 9 | 7
Completed | 11 | 6 | 4
Not Completed | 5 | 3 | 3
Not completed — Other | 2 | 0 | 0
Not completed — No longer met eligibility criteria | 2 | 2 | 0
Not completed — Unwilling to participate in study | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants in the treatment period (including titration phase and maintenance phase) who received at least 1 dose of ALO-02. This study was single-arm and data was reported by 3 arms to show dose related differences. The results were combined, not separated by 2 phases, due to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALO-02 <=20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg | Total
Number analyzed (Participants) | 16 | 9 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.0) | 15.2 (1.3) | 15.3 (1.1) | 14.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 12 | 5 | 2 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 6 | 5 | 26
  Black | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Steady-state Concentration (Css, av) of Oxycodone
Description: ALO-02 capsules consist of controlled-release pellets containing oxycodone hydrochloride (HCl) and naltrexone HCl. Oxycodone is a main component of this product.
Time Frame: Visit 4 (Day 21,28,35 or 42) or Visit 5 if not collected at Visit 4 (early termination or end of study, which occurred on Day 35,42,49 or 56) in Maintenance Phase
Population: The PK samples were collected but not analyzed and discarded due to early termination of the study.
Groups:
- ALO-02 <= 20 mg: Oral ALO-02 capsules average daily dose ≤ 20 mg BID (the average daily dose is the total dose amount divided by the total treatment days)
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Apparent Oral Clearance (CL/F) of Oxycodone
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK samples were collected but not analyzed and discarded due to early termination of the study.
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants With All-causality and Treatment-related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. All-causality AEs refer to any AE occurrence which needed not necessarily have a causal relationship with the treatment or usage. Treatment-related AEs refer to AEs that have a causal relationship with the treatment or usage. The majority of AEs were of mild to moderate severity.
Time Frame: Baseline up to Day 63
Population: The safety population consisted of all subjects who participated in the treatment period and received at least 1 dose of ALO-02.
Measure: Count of Participants; unit: Participants
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 16 | 9 | 7
Participants
  All-causality AEs | 14 | 8 | 7
  Treatment-related AEs | 9 | 6 | 6

4. Primary Outcome: Number of All-causality and Treatment-related AEs, by Intensity
Description: as for outcome 3
Time Frame: Baseline up to Day 63
Population: as for outcome 3
Measure: Number; unit: Events
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 16 | 9 | 7
Events
  All-causality AEs (mild) | 38 | 32 | 26
  All-causality AEs (moderate) | 15 | 10 | 12
  All-causality AEs (severe) | 0 | 0 | 3
  Treatment-related AEs (mild) | 19 | 24 | 16
  Treatment-related AEs (moderate) | 6 | 4 | 6
  Treatment-related AEs (severe) | 0 | 0 | 0

5. Primary Outcome: Number of Participants With All-causality and Treatment-related Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. All-causality SAEs refer to any SAE occurrence which needed not necessarily have a causal relationship with the treatment or usage. Treatment-related SAEs refer to SAEs that have a causal relationship with the treatment or usage.
Time Frame: Baseline up to Day 63
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 16 | 9 | 7
Participants
  All-causality | 0 | 0 | 2
  Treatment-related | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS)
Description: The COWS contains 11 common opiate withdrawal signs or symptoms rated by the clinician.The summed score of the 11 items is used to assess a subject's level of withdrawal. A subject assessed with a COWS score>= 13 was treated for opiate withdrawal signs and symptoms according to the investigator's medical judgment. The total COWS score ranges from 0 to 48. Higher scores indicate worse outcome. Different score ranges represent different severities of withdrawal: no withdrawal (<5), mild (5-12), moderate (13-24), moderately severe (25-36), and severe (>36)
Time Frame: Screening, Day 1, Titration Phase: Weeks 1,2,3,4; end of titration phase; Maintenance phase: Weeks 2, 4; early termination at titration phase, end of maintenance phase.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 16 | 9 | 7
Participants
  COWS score<5 (screening) | 15 | 9 | 7
  COWS score 5-12 (mild) (screening) | 1 | 0 | 0
  COWS score<5 (end of maintenance phase) | 15 | 8 | 7
  COWS score 5-12 (mild) (end of maintenance phase) | 1 | 1 | 0

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Oxycodone
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK samples were collected but not analyzed and discarded due to early termination of the study.
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Systemic Exposure Levels of the Metabolites of Oxycodone (Oxymorphone and Noroxycodone), Naltrexone, and 6-β-naltrexol.
Description: Oxymorphone and noroxycodone are major metabolites of Oxycodone and 6-β-naltrexol is the major metabolite of naltrexol.
Time Frame: as for outcome 1
Population: The PK samples were collected but not analyzed and discarded due to early termination of the study.
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Maximum Changes in Vital Signs (Blood Pressure, Heart Rate, Respiratory Rate) Meeting Categorical Summarization Criteria
Description: Following parameters were analyzed for examinations of vital signs: resting systolic and diastolic blood pressure, heart rate, and respiratory rate. In this study, there were only participants meeting the maximum decrease from baseline in systolic blood pressure (SBP) >= 30 mmHg and diastolic blood pressure (DBP) >=20 mmHg criteria. None of the vital sign changes were clinically significant.
Time Frame: Baseline up to Day 58
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 16 | 9 | 7
Participants
  Maximum decrease from baseline in SBP>=30mmHg | 1 | 0 | 1
  Maximum decrease from baseline in DBP>=20mmHg | 1 | 2 | 0

10. Secondary Outcome: Number of Participants With Laboratory (Lab) Abnormalities (Hematology and Chemistry)
Description: Following parameters were analyzed for hematologic laboratory tests: hemoglobin, hematocrit, red blood cells, mean corpuscular volume, platelets, white blood cells, lymphocytes (absolute & %), neutrophils (absolute & %), basophils (absolute & %), eosinophils (absolute &%), monocytes (absolute & %). Following parameters were analyzed for chemical laboratory tests: bilirubin,aspartate aminotransferase, alanine aminotransferase,alkaline phosphatase, protein(total), albumin,blood urea nitrogen, creatinine, cholesterol, sodium, potassium,chloride, calcium, phosphate, bicarbonate, glucose, creatine kinase. None of the lab abnormalities were clinically significant.
Time Frame: Baseline up to Day 77
Population: The laboratory data analysis set included only those participants who had post baseline lab results.
Measure: Count of Participants; unit: Participants
Arm/Group | ALO-02 <= 20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
Number analyzed (Participants) | 15 | 9 | 7
Participants
  Hematology | 8 | 5 | 4
  Chemistry | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Day 63
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | ALO-02 <=20 mg | ALO-02 >20-40 mg | ALO-02 >40-80 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9 | 2/7
Other Adverse Events (participants affected / at risk) | 14/16 | 8/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALO-02 <=20 mg (N=16) | ALO-02 >20-40 mg (N=9) | ALO-02 >40-80 mg (N=7)
Migraine (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ALO-02 <=20 mg (N=16) | ALO-02 >20-40 mg (N=9) | ALO-02 >40-80 mg (N=7)
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 1
Miosis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 2
Nausea (Gastrointestinal disorders) | 5 | 4 | 2
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 0 | 1
Feeling of body temperature change (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0/4 | 0/4 | 1/5
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 — This event occurred on Study Day -2 and should be included in medical history instead of AE section. The error was not identified until after database lock.
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 2
Dizziness exertional (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 3 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Social anxiety disorder (Psychiatric disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor's decision instead of safety or efficacy reasons. Early termination led to small numbers of participants summarized or described and PK samples were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results

DOCUMENTS (2):
  • Study Protocol (2006-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT02680847/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT02680847/SAP_001.pdf